CLINICAL TRIAL: NCT00926627
Title: A Prospective Randomized, Double Blind, Placebo-controlled, Safety and Efficacy Study of Bosentan as add-on Therapy in Progressive Pulmonary Sarcoidosis
Brief Title: Safety and Efficacy Study of Bosentan in Progressive Pulmonary Sarcoidosis
Acronym: BOPSAC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Not enough patients with the specified criteria could not
Sponsor: Daniel Doberer (Other)
Responsible Party: Sponsor-Investigator, Daniel Doberer, Research Associate, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT - 2007-005117-18
Record Dates: First submitted 2009-06-22; First posted 2009-06-23 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Sarcoidosis; Pulmonary Hypertension
Keywords: endothelin receptor antagonist; bosentan
MeSH Terms: conditions — Sarcoidosis; Hypertension, Pulmonary | interventions — Bosentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): placebo b.i.d.
  Interventions: Drug: placebo
- Bosentan (Experimental): 62.5 mg/125 mg bosentan b.i.d.
  Interventions: Drug: bosentan

INTERVENTIONS:
Drug: bosentan — 62.5 mg tablets b.i.d. administered orally for 4 weeks followed by the maintenance dose of 125 mg b.i.d. (62.5 mg b.i.d. if body weight < 40 kg/90 lb)
  Arms: Bosentan
Drug: placebo — identical preparation as the study drug, but without the active substance, administered b.i.d.
  Arms: Placebo

SUMMARY:
Progressive pulmonary sarcoidosis occurs in up to twenty percent of patients who require persistent treatment, but available treatment options have shown considerable long-term toxicity and uncertain or unproven efficacy. In these patients, pulmonary fibrosis and pulmonary hypertension are common complications which have major prognostic impact. Endothelin-1 (ET-1) has been demonstrated to play a key role in pulmonary fibrosis and pulmonary hypertension, and a potential role in pulmonary sarcoidosis. ET-1 is a potent vasoconstrictor and can promote fibrosis, cell proliferation, and remodeling, and is pro-inflammatory. Preliminary data have shown the therapeutic potential of the endothelin receptor antagonist (ERA) bosentan in sarcoidosis associated pulmonary hypertension.

In this light, the therapeutic potential of bosentan as an add-on treatment in progressive pulmonary sarcoidosis needs to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure.
* Male and female patients aged > 18 and < 70 years.
* Histologically proven sarcoidosis diagnosed at least one year before screening.
* Diagnosis of sarcoidosis and with evidence of pulmonary parenchymal disease on chest X-ray or CT (radiological stage II, III) with or without pulmonary hypertension. Subjects with concurrent extrapulmonary sarcoidosis are encouraged to be enrolled.
* Progressive disease, defined as follows:

  * Deterioration in the 3-12 month period prior to screening in at least two of the following criteria:

    * increase in clinical symptoms (cough, shortness of breath, chest pain, fatigue or hemoptysis).
    * lung function: decrease of 10% in TLC, FVC or DLCO.
    * worsening of radiographic opacities.
  * Have been receiving pre-study treatment with prednisolone (or equivalent dose of corticosteroid) as a single agent (≥ 10 mg/day) or other immunosuppressants (methotrexate, azathioprine, cyclophosphamide, TNF inhibitors, etc.) within the 3-month period immediately prior to screening. Patients must be on a stable dose of these medications for > 4 weeks before starting the study medication.
* AST and ALT values within three times upper limit of normal.
* Ability to communicate well with the investigator, in the local language, and to understand and comply with the requirements of the study.
* Negative pregnancy test in female patients.
* Adequate contraception in female patients of childbearing age.

Exclusion Criteria:

* Known hypersensitivity to any excipients of the drug formulation or to bosentan.
* Treatment with another investigational drug within 3 months prior to screening.
* Pulmonary sarcoidosis:

  * without disease progression as defined above
  * with radiological stage I
  * with radiological stage IV (pulmonary fibrosis with evidence of honey-combing, hilar retraction, bullae and cysts)
* Other cause of pulmonary disease:

  * Active tuberculosis (or positive Quantiferon test), fungi infection, lymphoma.
  * Chronic obstructive pulmonary disease, asthma, interstitial lung disease other than sarcoid-related
* Anamnesis of beryllium or asbestos exposition
* Previous smoking (> 10 PY), or active smoker
* Previous administration of bosentan
* Positive results from the hepatitis serology, except for vaccinated subjects, at screening.
* Positive results from the HIV serology at screening.
* Malignancy requiring chemotherapy or radiation
* Uncontrolled other disease like

  * Chronic heart failure (NYHA III, IV)
  * Diabetes mellitus (blood glucose 2x per day > 250 mg/dl , HbA1c > 10 %)
  * Arterial hypertension (SBP > 180 mmHg)
* Concomitant treatment with cyclosporine A
* Concomitant treatment with tacrolimus or sirolimus
* Concomitant treatment with glibenclamide
* Are pregnant, nursing, or planning pregnancy during the trial or within six month period thereafter.
* Have a known substance dependency (drug or alcohol within 3 years of screening).
* Presumed non-compliance.
* Legal incapacity or limited legal capacity at screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Treatment efficacy is assessed by a composite clinical score, including six parameters: Pulmonary function test (FVC and DLCO), Blood gas analysis (AaDO2), HRCT (Oberstein score), 6 minute walk test (6-MWD), Dyspnoea (ATS dyspnea scale) | 6 months

SECONDARY OUTCOMES:
Assess safety and tolerability of bosentan in progressive pulmonary sarcoidosis | 6 months
To evaluate the efficacy of bosentan treatment in the subgroups of patents with and without sarcoidosis-associated pulmonary hypertension. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Doberer, MD, MSc, Study Director — Medical University of Vienna
Locations (2):
- Austria (2):
  - General Hospital Vienna, Vienna, Vienna
  - Wilhelminenspital Wien, Vienna, Vienna

REFERENCES:
- See also: Department of Clinical Pharmacology of the Medical University of Vienna — http://www.meduniwien.ac.at/klpharm/